CLINICAL TRIAL: NCT03012360
Title: Antimicrobial Treatment in Patients With Ventilator-associated Tracheobronchitis: a Prospective Randomized Placebo-controlled Double-blind Multicenter Trial
Brief Title: Antimicrobial Treatment in Patients With Ventilator-associated Tracheobronchitis
Acronym: TAVeM2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of inclusion pandemic, investigator reluctance, lower than expected incidence of infection
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015_66; 2016-000735-41 (EudraCT Number)
Record Dates: First submitted 2016-12-13; First posted 2017-01-06 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Mechanical Ventilation Complication; Critical Illness
Keywords: Infectiology; Biology of infectious agents; Hygiene; Pneumology; Critical Care
MeSH Terms: conditions — Critical Illness | interventions — Ceftriaxone; Ciprofloxacin; Imipenem; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no antibiotic treatment for VAT (Placebo Comparator): 3 days of placebo
  Interventions: Drug: placebo
- antibiotic treatment for 3 days (Experimental): Patients randomized in one of the two experimental groups will receive 3 days of antimicrobials. Antibiotic treatment is standardized, based on the time of onset of VAT, and presence of risk factors for MDR bacteria:
  * patients with early-onset VAT (< 5 days of mechanical ventilation), with no risk factor for MDR will receive ceftriaxone .
  * patients with late-onset VAT (≥5 days of mechanical ventilation), or with at least one risk factor for multidrug resistant bacteria will receive imipenem , and ciprofloxacin as empirical treatment.
  When methicillin-resistant Staphylococcus aureus (MRSA) is suspected linezolid will be added to empirical treatment.
  3 days of imipenem and ciprofloxacin with optional linezolid, followed by 4 d of placebo
  Interventions: Drug: ceftriaxone; Drug: ciprofloxacin; Drug: imipenem; Drug: linezolid; Drug: placebo

INTERVENTIONS:
Drug: ceftriaxone — 2 g iv every 24h
  Arms: antibiotic treatment for 3 days
Drug: ciprofloxacin — 400 mg iv every 8h
  Arms: antibiotic treatment for 3 days
Drug: imipenem — 1 g iv every 8h
  Arms: antibiotic treatment for 3 days
Drug: linezolid — 600 mg iv every 12h
  Arms: antibiotic treatment for 3 days
Drug: placebo — The SSI 0.9% or dextrose 5% used are based on routine procedure in different participating centers.Placebo will be prepared using IV bags, with the same of quantity as IMP

SUMMARY:
Antimicrobial treatment could be beneficial in patients with ventilator-associated tracheobronchitis (VAT). The hypothesis of this study is that antibiotic treatment for VAT (3 or 7 days), compared with no antibiotic treatment, would reduce the incidence of transition from VAT to ventilator-associated pneumonia (VAP).

DETAILED DESCRIPTION:
The main objective of this randomized controlled multicenter double-blind trial is to assess the efficiency of two durations (3 or 7 days) of antibiotic treatment for VAT, compared with no antibiotic treatment, in reducing the incidence of transition from VAT to ventilator-associated pneumonia (VAP).

Secondary objectives are to determine the impact of two durations (3 or 7 days) of antibiotic treatment for VAT, compared with no antibiotic treatment, on:

* duration of mechanical-ventilation free days
* duration of antibiotic free days
* length of ICU stay
* mortality at day 28 and day 90
* incidence of ICU-acquired colonization related to multidrug resistant (MDR) bacteria
* incidence of ICU-acquired infection related to MDR bacteria
* incidence of ventilator-associated events After informed consent, patients will be randomized (1:1:1) to receive 0 (control group), 3 or 7 days (experimental groups) of antibiotic treatment for VAT

Antibiotic treatment is standardized, based on the time of onset of VAT, and presence of risk factors for MDR bacteria:

* patients with early-onset VAT with no risk factor for MDR bacteria will receive ceftriaxone (2 g iv every 24h).
* patients with late-onset VAT (after day 4 of mechanical ventilation), or with at least one risk factor for MDR bacteria will receive imipenem (1 g iv every 8h), and ciprofloxacin (400 mg iv every 8h) as empirical treatment. When methicillin-resistant Staphylococcus aureus is suspected, linezolid (600 mg iv every 12h) will be added to empirical treatment.

Patients randomized in control group will receive 7 days of placebo, and those randomized in the first experimental arm (3 days of antibiotics) will receive 4 days of placebo.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients hospitalized in the ICU with a first episode of VAT diagnosed >48 hours after starting invasive mechanical ventilation are eligible for this study.

VAT is defined using the following criteria:

1. absence of new infiltrate on chest X ray
2. two of the three following conditions: fever > 38.5 °C or <36.5, leucocyte count > than 12 000 cells per μL or <than 4000 cells per μL purulent tracheal secretions
3. and positive tracheal aspirate (≥105 cfu/mL)

Exclusion Criteria:

* long-term tracheostomy at ICU admission
* patients who develop VAP before VAT
* patients already receiving antibiotics active against all the microorganisms responsible for VAT
* severe immunosuppression
* pregnancy or breastfeeding
* patients <18 years
* patients already included in another study, with potential interaction with the primary objective of the current study
* known resistance to imipenem and ciprofloxacin of bacteria responsible for VAT
* treatment limitation decisions
* moribund patients (likely to die within 24 h)
* allergy to any of study drugs: hypersensitivity to any carbapenem, severe hypersensitivity (for example anaphylactic reaction or severe cutaneous reaction) to any other antibiotic form beta-lactam group (such as penicillin or cephalosporin), severe hypersensitivity (for example anaphylactic reaction) to any other antibiotic from beta-lactam group (penicillin, monobactam or carbapenem), hypersensitivity to quinolones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with a transition from VAT to VAP, | from randomization to day 28 (4 weeks)
  VAP is defined using the following criteria:
  1. new or progressive pulmonary infiltrate
  2. two of the following criteria: temperature >38°C or <36.5°C leukocyte count >12,000/μL or <4,000/μL purulent endotracheal aspirate
  3. positive tracheal aspirate (≥105 cfu/mL) or bronchoalveolar lavage (≥104 cfu/mL).
  VAP will be considered as subsequent to VAT, when it is diagnosed >24h after VAT occurrence. Only first episodes of VAP diagnosed >48h after starting mechanical ventilation will be taken into account.

SECONDARY OUTCOMES:
duration of mechanical ventilation-free days | from randomization to day 28 (4 weeks)
duration of antibiotic free-days | from randomization to day 28 (4 weeks)
length of ICU stay | from randomization to day 28 (4 weeks)
mortality | at day 28 and day 90 after randomization
percentage of patients with ICU-acquired colonization related to MDR bacteria | from randomization to day 28 (4 weeks)
percentage of patients with ventilator-associated events | from randomization to day 28 (4 weeks)
percentage of patients with ICU-acquired infection related to MDR bacteria | from randomization to day 28 (4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Saad NSEIR, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No